CLINICAL TRIAL: NCT06629415
Title: Intravenous Injection Versus Transhepatic Intracholecystic Injection of Indocyanine Green (ICG) to Outline Biliary Tree During Laparoscopic Cholecystectomy
Brief Title: Using Indocyanine Green (ICG) to Outline Biliary Tree During Laparoscopic Cholecystectomy
Acronym: ICG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mahmoud Rady, Researcher, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PT (657)
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Calculous Cholecystitis; Laparoscopic Cholecystectomy
Keywords: common bile duct injury, Intracholecystic, fluorescence cholangiography, indocyanine green, laparoscopic cholecystectomy.
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous Injection Injection of Indocyanine Green (ICG) (Active Comparator): 7.5 mg (3 ml of a 25 mg/10 ml solution) of indocyanine green was injected intravenously in the pre-operative holding area at least 20 minutes before surgery to outline the biliary tree during laparoscopic cholecystectomy.
  Interventions: Drug: Indocyanine Green
- Transhepatic intracholecystic injection of Indocyanine Green (ICG) (Active Comparator): Intracholecystic injection of ICG was done in 30 patients. Twenty 1.25 mg particles, one from a 25 mg ICG vial, were separated under aseptic conditions.
  Interventions: Drug: Indocyanine Green Drug

INTERVENTIONS:
Drug: Indocyanine Green — injecting 7.5 mg (3 ml of a 25 mg/10 ml solution) intravenously in the pre-operative holding area at least 20 minutes before surgery.
  Before dissecting the adhesions surrounding the hepatoduodenal ligament, fluorescence cholangiography (FC) is carried out to determine the anatomy of the extrahepatic bile ducts by converting the full-color images to fluorescence images using filter switches on the camera head and/or light source in the laparoscopic imaging system (Fig. 1). The "critical view of safety" is then reached by dissecting Calot's triangle and using FC to verify whether the accessory bile ducts are present or absent throughout the procedures. It is necessary to acquire fluorescence image
  Arms: Intravenous Injection Injection of Indocyanine Green (ICG)
Drug: Indocyanine Green Drug — 1.25 mg of ICG powder was dissolved in 3 cm of saline, and the concentration was roughly 0.04 mg after each 1 cm of saline was diluted by 9 cm of saline. In order to prevent dye leakage that might result in false FC results, a veress needle was inserted through the abdominal wall and into the gall bladder fundus through the liver bed. The puncture site was then cauterized.
  Arms: Transhepatic intracholecystic injection of Indocyanine Green (ICG)

SUMMARY:
The current study shows that Indocyanine green (ICG)-fluorescence cholangiography can be useful in identifying the extrahepatic biliary anatomy during Calot's triangle dissection. By avoiding hepatic fluorescence, the transhepatic intracholecystic-ICG route can increase the bile duct-to-liver contrast with less expense and no risk of hypersensitivity reactions than the intravenous ICG injection method. We recommend to use both techniques in case of acute cholecystitis with cystic duct obstruction. In cases of liver cirrhosis, we recommend transhepatic IC-ICG as IV-ICG is limited.

DETAILED DESCRIPTION:
Materials and Methods After informed consent, 60 patients with acute or chronic cholecystitis scheduled for NIR-ICG fluorescent cholangiography during LC were consecutively included in the study. ICG was ad ministered intravenously or intracholecystic injection during surgery. This prospective randomized comparative was evaluated based mainly on the clear anatomical delineation of the gall bladder, cystic duct, hepatic ducts and common bile duct. This study had been conducted from 2022 to 2024 with the approval of the institutional ethics committee.

Inclusion criteria included patients from 16 to 80 years old, patients with gall bladder pathology (cholecystitis, gall bladder polyp) and patients fit for laparoscopic cholecystectomy.

Exclusion criteria included patients with contraindication for laparoscopic cholecystectomy (for example patients had significant pulmonary or cardiac problems or severe renal insufficiency), intraoperative dye spillage during dissection of the gallbladder, obstructive jaundice, proven or suspected allergies to ICG, pregnancy or lactation.

The patients were classified into 2 groups, group A patients (n = 30) were chosen for intravenous injection of ICG while group B patients (n = 30) were chosen for transhepatic intracholecystic injection of ICG during cholecystectomy.

To randomise, a sealed opaque envelope was chosen based on a computer-generated random sequence. Surgeons with extensive experience in biliary surgery performed all laparoscopic procedures. The patients age, sex, BMI, comorbidities, and cholecystectomy indication were among their characteristics. Perioperative data included the percentage of non-elective versus elective procedures, the length of time from skin incision to skin closure during the procedure, the location of intraoperative drains, the estimated blood loss (EBL), and the necessity of switching from a laparoscopic to an open approach.

Of note, patients undergoing a concomitant procedure during LC (i.e., esophagogastroduodenoscopy, liver biopsy, lap gastric band removal, etc.) were excluded from the operative time analysis.

A laparoscopic system was used in each and every instance. The image is created by a top-of-the-line full-HD camera system that is mounted to a laparoscope with a 30° field of view and a 10mm diameter. It was equipped with a unique filter for the best detection of NIR fluorescence and white light without the need for manual switching. The strong xenon light source provided excitation light for both the visible and NIR spectrums. The surgeon controled the changeover from conventional light to near-infrared light with a pedal. An expert image improvement system that allowed surgeons to select their preferred adjustable visualization modalities.

Thirty patients received intravenous ICG in group A (IV-ICG). In order to administer ICG, the standard protocol called for injecting 7.5 mg (3 ml of a 25 mg/10 ml solution) intravenously in the pre-operative holding area at least 20 minutes before surgery. Just before injection, a 25 mg vial of Indocyanine Green for Injection.

Before dissecting the adhesions surrounding the hepatoduodenal ligament, fluorescence cholangiography (FC) is carried out to determine the anatomy of the extrahepatic bile ducts by converting the full-color images to fluorescence images using filter switches on the camera head and/or light source in the laparoscopic imaging system. The "critical view of safety" was then reached by dissecting Calot's triangle and using FC to verify whether the accessory bile ducts are present or absent throughout the procedures. It was necessary to acquire fluorescence images of the bile ducts from both the ventral and dorsal sides of Calot's triangle. After confirming that there were no fluorescing structures other than the cystic duct (CD) connecting the gallbladder and the common hepatic duct (CHD), the CD was finally closed and divided.

In group B (IC-ICG): Transhepatic intracholecystic injection of ICG was done in 30 patients. 1.25 mg of ICG powder from a 25 mg ICG vial were separated under aseptic conditions and dissolved in 3 ml of saline, and the concentration was roughly 0.04 mg after each 1 ml was diluted by 9 ml of saline. In order to prevent dye leakage that might result in false FC results, a veress needle was inserted through the abdominal wall and into the gall bladder fundus through the liver parenchyma (transhepatic), Then puncture site was cauterized. Then the same technique and images were taken as in group A.

Usually, the gallbladder was removed through the umbilical or epigastric port. From the moment the first incision was made until the last wound was closed, the operating time was tracked. On the first postoperative day, patients were sent home. An analysis was conducted on the following factors: operation time, dye spillage due to technique due to injection, cystic duct, common hepatic duct, common bile duct delineation, drain insertion, postoperative hospital stays, complications, and biliary injury.

Statistical methods Student's t test was used to compare the data with a normal distribution and the continuous variable data, which were provided as mean ± standard deviation. When appropriate, the Fisher's exact test or the Chi-square test were used to compare categorical variables, and logistic regression was employed for univariate analysis. SPSS version 20.0 was used for the statistical analysis (SPSS Inc., Chicago, IL, USA). P values less than 0.05 were regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of gall bladder pathology (cholecystitis, gall bladder polyp) Patients fit for laparoscopic cholecystectomy.

Exclusion Criteria:

Patients with contraindication for laparoscopic cholecystectomy (for example patients had significant pulmonary or cardiac problems or severe renal insufficiency).

Proven or suspected allergies to ICG. pregnancy or lactation.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
The rate of better delineation of the biliary tree during laparoscopic cholecystectomy | intraoperative and 2 weeks postoperative
  To detect the safety, efficacy, feasibility and accuracy in defining the biliary anatomy during laparoscopic cholecystectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
the data will be shared upon request from the principle investigator

REFERENCES:
- [Background] van Manen L, Handgraaf HJM, Diana M, Dijkstra J, Ishizawa T, Vahrmeijer AL, Mieog JSD. A practical guide for the use of indocyanine green and methylene blue in fluorescence-guided abdominal surgery. J Surg Oncol. 2018 Aug;118(2):283-300. doi: 10.1002/jso.25105. Epub 2018 Jun 24. PMID 29938401